CLINICAL TRIAL: NCT00234195
Title: A Pilot Study of the Efficacy and Tolerability of Bupropion Extended Release (Wellbutrin XL) for the Treatment of Major Depressive Disorder in Women With Breast Cancer
Brief Title: Wellbutrin XL, Major Depressive Disorder and Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prot105042; 29000-J08101
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer; Major Depressive Disorder
Keywords: Breast Cancer; Major Depressive Disorder
MeSH Terms: conditions — Breast Neoplasms; Depressive Disorder, Major | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bupropion extended release (Wellbutrin XL)

SUMMARY:
* To evaluate the efficacy of bupropion extended release (Wellbutrin XL™) in the treatment of Major Depressive Disorder in women with breast cancer.
* To evaluate the tolerability of bupropion extended-release (Wellbutrin XL™) in these patients

DETAILED DESCRIPTION:
This is research study for women diagnosed with breast cancer and major depression. Women with breast cancer who are depressed may report greater pain, poorer quality of life and worse overall functioning than those without depression. The study will determine whether or not bupropion extended release (Wellbutrin XLTM) is useful in lessening the symptoms of depression in women with breast cancer. One reason for conducting this research with bupropion extended release (Wellbutrin XLTM) instead of another antidepressant is because bupropion has a lower likelihood of causing the side effects of weight gain, sexual dysfunction, and fatigue, which may be important for women with breast cancer and may even have a beneficial effect on these symptoms.

Bupropion extended release (Wellbutrin XL™)is approved by the United States Food and Drug Administration (FDA) for the treatment of major depression.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Diagnosis of breast cancer, confirmed by histopathology; Stages 0, I, II, IIIA, or IIIB
* Clinical diagnosis of Major Depressive Disorder (DSM-IV-TR)
* Hospital Anxiety and Depression Scale (Zigmond and Snaith, 1983) depression subscale score of 11 or greater
* Montgomery Asberg Depression Rating Scale (MADRS; Montgomery and Asberg, 1979) score of 25 or greater at Screening and Baseline visits
* Use of antidepressants in a previous episode of major depression or in the past for any other indication does not affect the patient's inclusion in this study.
* During the current episode of major depressive disorder, as stated in the Exclusion criteria, failure to respond to one or more adequate trials of an antidepressant will exclude the patient from the study since this is not a study of "treatment-resistant depression".
* During the study, the patient may not use any other antidepressants.

Exclusion Criteria:

* Presence of another current clinically significant Axis I disorder like bipolar disorder, schizophrenia, or panic disorder
* Current (in past 6 months) comorbid active substance abuse or dependence
* Failure to respond to one or more adequate trials of an antidepressant in the current episode of MDD
* A reduction in MADRS score of 20% or greater from Screening to Baseline visit
* Clinically significant laboratory abnormalities that in the judgment of the Investigator would increase risk of adverse effects with bupropion
* Pregnant or lactating women
* History of an eating disorder, seizures, head injury, or other intracranial pathology because these conditions are usually contraindications to the use of bupropion XL
* Previous allergy or intolerance to bupropion
* Patients judged to be at significant suicidal risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of bupropion extended release (Wellbutrin XL™) in the treatment of Major Depressive Disorder in women with breast cancer.
To evaluate the tolerability of bupropion extended-release (Wellbutrin XL™) in these patients

SECONDARY OUTCOMES:
To evaluate the effect of bupropion extended-release (Wellbutrin XL™) on fatigue, sexual functioning, and pain in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mago, MD, Principal Investigator — Thomas Jefferson University Department of Psychiatry and Human Behavior
Locations (1):
- Thomas Jefferson University, Department of Psychiatry, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619